CLINICAL TRIAL: NCT03321578
Title: National Infection Trainees Collaborative for Audit and Research (NITCAR) Service Evaluation: The Prevalence, Aetiology and Management of Hospital-onset Diarrhoea on Medical, Surgical and Elderly Care Wards in the NHS
Brief Title: Hospital Onset Diarrhoea Investigation
Acronym: HOODINI
Status: Completed | Type: Observational
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Collaborators: Aneurin Bevan University Health Board (Other); Northern Health and Social Care Trust (Other Government); Barnsley Hospital NHS Foundation Trust (Other); Cambridge University Hospitals NHS Foundation Trust (Other); East Lancashire Hospitals NHS Trust (Other); Guy's and St Thomas' NHS Foundation Trust (Other); Hampshire Hospitals NHS Foundation Trust (Other); Harrogate & District NHS Foundation Trust (Other); Hull University Teaching Hospitals NHS Trust (Other Government); Mid Yorkshire Teaching NHS Trust (Other); NHS Greater Glasgow and Clyde (Other); NHS Lothian (Other Government); Nottingham University Hospitals NHS Trust (Other); Oxford University Hospitals NHS Trust (Other); Papworth Hospital NHS Foundation Trust (Other Government); Sheffield Teaching Hospitals NHS Foundation Trust (Other); South Tees Hospitals NHS Foundation Trust (Other); Royal Free Hospital NHS Foundation Trust (Other); The Royal Wolverhampton Hospitals NHS Trust (Other Government); Torbay and South Devon NHS Foundation Trust (Other); South Eastern Health and Social Care Trust (Other); University Hospitals Coventry and Warwickshire NHS Trust (Other); George Eliot Hospital NHS Trust (Other); University Hospitals, Leicester (Other); York Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: v10.5
Record Dates: First submitted 2017-10-23; First posted 2017-10-25 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Diarrhea
Keywords: nosocomial; hospital acquired; clostridium difficile
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This service evaulation aims to investigate how common diarrhoea is in hospital patients on medical, surgical and elderly care wards, what it is due to and how it is managed.

DETAILED DESCRIPTION:
Latest National Health Service (NHS) England guidelines for the assessment of Clostridium difficile infection (CDI) cases recommend that acute hospitals collect data on the prevalence of hospital-onset diarrhoea in their organisations, and how it is managed, including if patients are appropriately tested for CDI.

The aims of this multi-centre service evaluation are therefore to:

* Determine the prevalence of hospital-onset diarrhoea on adult medical, surgical and care of the elderly wards in the NHS
* Investigate how hospital-onset diarrhoea is managed, including whether patients are tested for CDI according to Department of Health (DoH) England standards
* Investigate the aetiology of hospital-onset diarrhoea on adult medical, surgical and care of the elderly wards in the NHS, based on previously described causes

Data will be collected at participating centres on two days, one between 11-15/Jan/2016 and one between 6-10/Jun/2016. Hospitals will be able to choose locally which two days. On those days investigators from the local Microbiology and/or Infection Prevention teams will screen all patients on pre-identified wards, who have been admitted for ≥72 hours, for hospital-onset diarrhoea. For all patients that meet the definition of hospital-onset diarrhoea their medical notes and charts will be reviewed, to ascertain potential causes and how they have been managed.

This service evaluation should help participating hospitals to investigate hospital-onset diarrhoea in their own institutions, as well as generating a dataset that is representative of the problem across the NHS, and therefore of use to other centres.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to hospital for ≥72 hours at the time of data collection for the service evaluation
* Presence of hospital-onset diarrhoea (defined as ≥ 2 episodes of unformed stools (Bristol Stool Chart type 5-7) during the day before the service evaluation, with the onset of the diarrhoea being more than 48 hours after admission to hospital)

Exclusion Criteria:

* Patients admitted to the ward for ≤72hour at the time of data collection for the service evaluation
* Patients with diarrhoea since admission or in whom it developed within the first 48 hours of admission
* Patients receiving end of life care

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cases (patients with hospital-onset diarrhoea)
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Point-prevalence of hospital-onset diarrhoea | At enrollment

SECONDARY OUTCOMES:
• The proportion of patients with hospital-onset diarrhoea who have been assessed for the problem by a member of the clinical team. | At enrollment
• The proportion of patients with hospital-onset diarrhoea that are tested for CDI (both overall and amongst those who do and do not have an alternative explanation for the diarrhoea). | Up to 72 hours after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kirby, MBBS, Study Director — Leeds Teaching Hospitals NHS Trust; Jonathan AT Sandoe, MBChB, Study Director — Leeds Teaching Hospitals NHS Trust
Locations (24):
- United Kingdom (24):
  - Antrim Area Hospital (Northern Health and Social Care Trust), Antrim
  - Barnsley Hospital NHS Foundation Trust, Barnsley
  - East Lancashire Hospitals NHS Trust, Blackburn
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - University Hospitals Coventry and Warwickshire + George Eliot Hospital NHS Trust, Coventry
  - Ulster Hospital (South Eastern Health and Social Care Trust), Dundonald
  - NHS Lothian and NHS Fife, Edinburgh
  - NHS Greater Glasgow and Clyde, Glasgow
  - Harrogate and District NHS Foundation Trust, Harrogate
  - Hull and East Yorkshire Hospitals NHS Trust, Hull
  - University Hospitals of Leicester NHS Trust, Leicester
  - Guy's & St Thomas' NHS Foundation Trust, London
  - The Royal Free London NHS Foundation Trust, London
  - South Tees Hospitals NHS Foundation Trust, Middlesbrough
  - Aneurin Bevan University Health Board, Newport
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford University Hospitals NHS Trust, Oxford
  - Papworth Hospital NHS Foundation Trust, Papworth Everard
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - Torbay and South Devon Healthcare NHS Foundation Trust, Torbay
  - Mid Yorkshire NHS Trust, Wakefield
  - Hampshire Hospitals NHS Foundation Trust, Winchester
  - The Royal Wolverhampton NHS Trust, Wolverhampton
  - York Teaching Hospital NHS Foundation Trust, York

IPD SHARING:
Plan to Share IPD: No